CLINICAL TRIAL: NCT03904680
Title: Studying the Effect of Methotrexate Alone Versus Methotrexate and Vitamin D on the Cardiovascular Risk of Psoriatic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Raafat Said, Lecturer of Dermatology Department, Faculty of Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Psoriasis
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Cardiovascular risk; Methotrexate; Vitamin D
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate; Vitamin D

STUDY DESIGN:
Intervention Model Description: The patients will be randomly divided into 2 groups:
  Group A: 15 patients will take methotrexate weekly for 3 months for the treatment of psoriasis.
  Group B: will take methotrexate weekly in addition to Vitamin D injections monthly for 3 months for treatment of psoriasis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methotrexate (Active Comparator): 15 patients will take methotrexate weekly with the dose of 0.2-0.5 mg/kg/week for 3 months.
  Interventions: Drug: Methotrexate
- Methotrexate and Vitamin D (Active Comparator): 15 patients will take methotrexate weekly with the dose of 0.2-0.5 mg/kg/week and Vitamin D intramuscular injections with the dose of 200,000 IU per month for 3 months.
  Interventions: Drug: Methotrexate; Drug: Vitamin D

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 2.5 mg tablet
Drug: Vitamin D — Vitamin D 200,000 IU ampules
  Arms: Methotrexate and Vitamin D

SUMMARY:
The prevalence of cardiovascular risk in psoriasis has been reported in previous studies.Various studies have also shown that systemic treatments for psoriasis, including methotrexate, may significantly decrease this cardiovascular risk. We proposed that the addition of vitamin D may not only improve the therapeutic effect of various treatment modalities but also increase its effect on decreasing the cardiovascular risk in psoriasis. So our aim of work is to assess the Clinical improvement and cardiovascular risks in psoriatic patients after treatment with methotrexate alone with the dose of 0.2-0.5 mg/kg/week for three months in comparison to combined methotrexate with the same dose and vitamin D injection with the dose of 200,000 IU per month for 3 months.

Each patient will do the following before starting treatment& after 3 months:

1. Fasting blood sugar, 2 hours postprandial and glycosylated hemoglobin
2. Liver and Kidney function tests.
3. Cardiovascular risk assessment by measuring the intima media thickness of carotid arteries using Carotid duplex and High sensitive C reactive protein measuring by particle-enhanced immunonephelometry on autoanalyzer.
4. Lipid profile (HDL, LDL, cholesterol and triglycerides).
5. Calculate body mass index and measure blood pressure
6. Albumin /creatinine ratio
7. Serum vitamin D level. Clinical response will be evaluated by Psoriasis Area and Severity index (PASI) & Psoriasis Disability Index (PDI) scores before and after 3 months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patient not on systemic treatment at least for 3 months before inclusion in the study
* PASI >10

Exclusion Criteria:

* Patients with autoimmune diseases.
* Patients with liver disease or kidney diseases
* Patients with Diabetes mellitus
* Females in child bearing period not using methods of contraception
* Any associated dermatological disease
* Evidence of infection
* Pregnancy and lactation
* Patients taking vitamin D

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change in Intima Media thickness of carotid arteries from baseline | Baseline and 12 weeks
  Intima Media thickness of left and right common carotid arteries, bulb of common carotid arteries and internal carotid arteries as measured by carotid duplex before starting the treatment and after 3 months of treatment.
Change in high sensitive C- Reactive protein from baseline | Baseline and 12 weeks
  Change in high sensitivity C-reactive protein (hsCRP), a soluble biomarker of systemic inflammation, after 3 months of treatment from baseline.
Psoriasis Area and Severity index change (PASI) | Baseline and 12 weeks
  Change in PASI after 3 months of treatment from baseline

REFERENCES:
- [Background] Furue M, Tsuji G, Chiba T, Kadono T. Cardiovascular and Metabolic Diseases Comorbid with Psoriasis: Beyond the Skin. Intern Med. 2017;56(13):1613-1619. doi: 10.2169/internalmedicine.56.8209. Epub 2017 Jul 1. PMID 28674347
- [Background] Fu LW, Vender R. Systemic role for vitamin d in the treatment of psoriasis and metabolic syndrome. Dermatol Res Pract. 2011;2011:276079. doi: 10.1155/2011/276079. Epub 2011 Jun 5. PMID 21747838
- [Background] Manolis AA, Manolis TA, Melita H, Manolis AS. Psoriasis and cardiovascular disease: the elusive link. Int Rev Immunol. 2019;38(1):33-54. doi: 10.1080/08830185.2018.1539084. Epub 2018 Nov 20. PMID 30457023